CLINICAL TRIAL: NCT05194852
Title: In Shoulder Adhesive Capsulitis, Ultrasound-guided Anterior Hydrodilatation in Rotator Interval is More Effective Than Posterior Approach: a Randomized Controlled Study
Brief Title: Ultrasound-guided Anterior Hydrodilatation in Shoulder Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Hassan Abu-Zaid, associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hydro1
Record Dates: First submitted 2021-12-02; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Shoulder Capsulitis
MeSH Terms: interventions — Adrenal Cortex Hormones; Sodium Chloride; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: the participants and outcome assessor didn't know the group classification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Active Comparator): Group I received ultrasound-guided hydrodilatation with corticosteroid, saline, and local anesthetic via posterior intra-articular approach
  Interventions: Procedure: ultrasound-guided posterior hydrodilatation; Drug: corticosteroid, saline, and local anesthetic; Other: guided stretching and strengthening exercise program
- group 2 (Experimental): group II received the same ultrasound-guided hydrodilatation via anterior rotator interval approach
  Interventions: Procedure: ultrasound-guided posterior hydrodilatation; Other: guided stretching and strengthening exercise program

INTERVENTIONS:
Procedure: ultrasound-guided posterior hydrodilatation — Group I was treated through posterior approach; The injection needle is introduced at the skin surface just lateral to the transducer and in an oblique lateral to medial direction. Group II was treated through anterior rotator interval approach. A 21-gauge needle is introduced into the rotator interval using an oblique path within the imaging plane of the transducer; from lateral to medial, the needle tip is imaged in real time throughout its passage from superficial to deep and is positioned in the biceps tendon sheath between the coracohumeral ligament above and biceps tendon below. Both groups were given the same guided stretching and strengthening exercise program
Drug: corticosteroid, saline, and local anesthetic — corticosteroid, saline, and local anesthetic
  Arms: group 1
Other: guided stretching and strengthening exercise program — guided stretching and strengthening exercise program

SUMMARY:
A prospective randomized controlled study among 60 consecutive adhesive capsulitis to compare between the ultrasound-guided anterior hydrodilatation in rotator interval and the posterior approach.

DETAILED DESCRIPTION:
patients was randomized into two equal groups. Group I received ultrasound-guided hydrodilatation with corticosteroid, saline, and local anesthetic via posterior intra-articular approach; group II received the same ultrasound-guided hydrodilatation via anterior rotator interval approach.

Both groups received guided stretching exercises for 3 months after injection. Baseline and 3 months evaluation of pain by visual analogue scale (VAS), shoulder pain and disability index (SPADI), and range of motion (ROM) had been recorded for all patients.

A statistical power analysis was performed after sample size estimation, based on data from the current study (N = 60), comparing group I to group II.

Qualitative data was expressed as numbers and percentages, and Chi-squared test, Quantitative data were expressed as mean and standard deviation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 35 to 60 years,
* patients who suffered pain and stiffness in only one shoulder, for 1 to 6 months
* patients who had restriction of passive motion.

Exclusion Criteria:

* patients with previous trauma,
* patients with neurological
* patients with endocrinal diseases
* patients with shoulder tumor
* patients with arthritis
* people who had received intra-articular shoulder injection within the last 6 months.
* Patients with tendon tear

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
visual analoge state | 3 months
  minimum value: 0 maximum value: 10 higher scores mean a worse outcome.
shoulder pain and disability index | 3 months
  minimum value: 0 maximum value: 100 higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided